CLINICAL TRIAL: NCT04949906
Title: A Real World Study of Yangxuenao Granules Reducing Bleeding Risk in Patients With Acute Ischemic Stroke Treated With Intravenous Thrombolysis
Brief Title: Study on Yangxue Nao Granules Reducing the Risk of Stroke
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019439
Record Dates: First submitted 2021-06-27; First posted 2021-07-02 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The experimental group: The application of raising serum brain granules
  Interventions: Drug: Raise serum brain granules
- The control group: No nourishing serum brain granules are used
  Interventions: Drug: No nourishing serum brain granules are used

INTERVENTIONS:
Drug: Raise serum brain granules — Should Yangseronao granules be used in patients undergoing intravenous thrombolysis for the diagnosis of acute ischemic stroke
  Groups: The experimental group
Drug: No nourishing serum brain granules are used — No nourishing serum brain granules are used
  Groups: The control group

SUMMARY:
Objective: To explore the effectiveness of raising serum nao granules in reducing the risk of bleeding in patients with acute ischemic stroke treated with intravenous thrombolysis in the real world

DETAILED DESCRIPTION:
Objective: To explore the effectiveness of raising serum nao granules in reducing the risk of bleeding in patients with acute ischemic stroke treated with intravenous thrombolysis in the real world Study Design. This study was a single center real world study. Through the review data, this study included in January 1, 2017 to September 30, 2019, see a doctor at Peking University third hospital neurology, emergency diagnosis of acute ischemic stroke, and venous thrombolysis in patients with a queue, on the basis of whether the application have serum brain particles are divided into a group and the control group, serum application parameters and nonparametric comparison, K-M curve and Cox regression model were used to evaluate the effectiveness of Yangxuenao granules in reducing bleeding conversion after intravenous thrombolysis by comparing the number of microbleeding, stroke severity score and modified Rankin score after 3 months follow-up with the weighted craniocerebral magnetic sensitivity imaging sequence reexamined within 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* A cohort of patients admitted to the Department of Emergency Neurology at Peking University Third Hospital on January 1, 2017 and admitted on September 30, 2019, who were diagnosed with acute ischemic stroke and underwent intravenous thrombolysis.

Exclusion Criteria:

* Patients who underwent intravenous thrombolysis but were confirmed to be apoplexy
* like by imaging and other clinical examinations; Incomplete craniocerebral MRI examination;
* Bridging endovascular therapy;
* The previous application of Yangxuenao granules or other drugs with similar effects;

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of patients admitted to the Department of Emergency Neurology at Peking University Third Hospital on January 1, 2017 and admitted on September 30, 2019, who were diagnosed with acute ischemic stroke and underwent intravenous thrombolysis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Microhemorrhage (CMB) of T2* sequence in MRI after thrombolysis | 1 day
  The number of CMB is an important imaging marker reflecting microvascular injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Yniversity Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No